CLINICAL TRIAL: NCT03077698
Title: A Phase 2, Single Arm, Two Period Study of Sodium Cridanimod in Conjunction With Progestin Therapy in Patients With Endometrial Carcinoma
Brief Title: An Endometrial Cancer Study for Women With Recurrent or Persistent Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued due to a change in development strategy and not due safety concern.
Sponsor: Xenetic Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX-EC-2-02
Record Dates: First submitted 2017-02-27; First posted 2017-03-13 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Recurrent or persistent endometrial carcinoma; Progesterone Receptor Negative; Sodium Cridanimod
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — 10-carboxymethyl-9-acridanone; Estrogen Replacement Therapy; Megestrol Acetate

STUDY DESIGN:
Intervention Model Description: Phase 2, Single Arm, Two Period Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sodium Cridanimod & progestin therapy (Experimental): Sodium Cridanimod and progestin therapy (megestrol acetate) combination
  Interventions: Drug: Sodium Cridanimod; Drug: progestin therapy

INTERVENTIONS:
Drug: Sodium Cridanimod — The study will investigate the efficacy of Sodium Cridanimod in conjunction with progestin therapy in a population of subjects with endometrial cancer, who have failed progestin monotherapy or who have been identified as PrR negative.
Drug: progestin therapy — The study will investigator the use of progestin therapy in conjunction with Sodium Cridanimod
  Other Names: megestrol acetate

SUMMARY:
This is an open-label, multi-center, single-arm, two-period Phase 2 study. The study will investigate the efficacy of Sodium Cridanimod in conjunction with progestin therapy in a population of subjects with recurrent or persistent endometrial cancer, who have failed progestin monotherapy or who have been identified as Progesterone Receptor (PrR) negative. All patients must have endometrial cancer PrR status determined from an archival sample at Screening. The PrR status (positive or negative) will be determined by central laboratory by ImmunoHistoChemistry (IHC) testing.

There are two treatment periods and a follow-up period within the study.

DETAILED DESCRIPTION:
Treatment Period 1 (Progestin Monotherapy): During Treatment Period 1, all subjects determined to be PrR positive will receive progestin monotherapy, megestrol acetate, for up to 24 weeks. Subjects will have an MRI or CT scan after 12 and 24 weeks of progestin monotherapy, with response to treatment being assessed according to RECIST 1.1 criteria. All subjects that achieve disease control confirmed by tumor assessment after Treatment Period 1, will be ineligible to enter Treatment Period 2. These subjects will be terminated from the trial and treated according to local standards of practice, which may include continued progestin therapy.

Subjects determined to be PrR negative at Screening will not enroll into Treatment Period 1. These subjects will enroll directly into Treatment Period 2.

Treatment Period 2 (Combination Treatment): All subjects determined to be PrR negative at Screening and those who received at least 4 weeks of progestin monotherapy and who experienced disease progression at the conclusion of Treatment Period 1 will enter Treatment Period 2 of the study. During Treatment Period 2, subjects will receive Sodium Cridanimod in combination with continued progestin treatment, megestrol acetate. Subjects will receive treatment until disease progression as defined according to RECIST 1.1 criteria, with response assessments performed at 12-week intervals.

Follow-up Period: Once subjects progress during Treatment Period 2, they will return for a Safety Follow-up Visit 4 weeks following the last treatment, and then continue to be followed for an additional 12-month period for overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years of age or older;
2. Histologically confirmed serous carcinoma or endometrioid type of endometrial carcinoma (histological documentation of recurrence is not required);
3. Recurrent or persistent progressive disease which is refractory to curative therapy or established treatments and cannot be treated with surgery or radiotherapy;
4. Measurable disease, as defined by RECIST 1.1 criteria;
5. At least one "target lesion" to be used to assess response, as defined by RECIST 1.1 criteria. Tumors within a previously irradiated field will be designated as "non-target" lesions unless previous progression is documented;
6. Availability of archived tumor tissue sample that can be used for assessment of PrR status by the central laboratory;
7. GOG (Gynecologic Oncology Group) performance status 0-2 (refer to Appendix A);
8. Calculated Glomerular filtration rate ≥ 50 mL/min;
9. Total bilirubin ≤ 2.5 times upper limit of normal (ULN);
10. AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases);
11. Alkaline phosphatase ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver metastases);
12. Albumin ≥ 3.0 mg/dL;
13. Ability to take oral medication;
14. Patients able to understand the nature of the study and who are willing to give written informed consent;
15. And for Treatment Period 2 only: 1) Patients participating in Treatment Period 1 must have had disease progression after receiving at least 4 weeks of progestin therapy or 2) Patients must be determined as PrR negative status at Screening.

Exclusion Criteria:

1. Mixed histology of the tumor or evidence of tumor histology other than serous carcinoma or endometrioid type of endometrial carcinoma;
2. Concurrent systemic corticosteroid therapy;
3. Concurrent oral contraceptive use / Women of childbearing potential not using highly effective means of contraception;
4. Pregnancy confirmed by pregnancy test / Lactating women;
5. Prior therapy with hormonal progestin agents;
6. Patients who are candidates for treatment with standard chemotherapy agents (there is no limit to the number of lines of chemotherapy);
7. History of blood clot;
8. History of known bleeding disorder (i.e. disseminated intravascular coagulation or clotting factor deficiency);
9. Major surgery within 4 weeks prior to the start of the study;
10. Patients with clinically significant illnesses which, according to the Investigator, could compromise participation in the study;
11. History of other clinically active malignancies within 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma, or squamous carcinoma of the skin.
12. Known hypersensitivity or idiosyncratic reaction to any of the study drugs (Sodium Cridanimod, megestrol acetate, lidocaine) and excipients;
13. Patients with known brain metastases;
14. Patients currently receiving any other investigational agents;
15. Patients currently receiving any other anticancer therapies;
16. Participation in any other clinical study within the last 4 weeks prior to the start of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with endometrial cancer
Enrollment: 25 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Lockshin, PhD, Study Director — Xenetic Biosciences, Inc.
Locations (25):
- United States (25):
  - Providence St. Joseph Medical Center - Gynecology, Burbank, California
  - University of California - Irvine Healthcare, Irvine, California
  - UCLA, Los Angeles, California
  - St. Josephs Heritage Healthcare, Santa Rosa, California
  - University of Colorado School of Medicine, Division of Gynecologic Oncology, Aurora, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Northside Hospital [University Gynecologic Oncology], Atlanta, Georgia
  - MUMC - Curtis and Elizabeth Anderson Cancer Institute, Savannah, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - RUSH University Medical Center, Chicago, Illinois
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Women's Cancer Care [Mary Bird Cancer Center at Tammany Parish Hospital], Covington, Louisiana
  - St. Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute-UC Health Barrett Center, Cincinnati, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Magee Women's Hospital (UPMC), Pittsburgh, Pennsylvania
  - Rapid City Regional Cancer Care, Rapid City, South Dakota
  - UT Southwestern, Dallas, Texas
  - UT Galveston; University of Texas Medical Branch (UTMB), Galveston, Texas
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with PrR (+) tumors began in Treatment Period 1 receiving only Progestin Monotherapy. If PrR (+) subjects had disease progression they continued into Treatment Period 2 receiving Progestin and Sodium Cridanimod therapy. Subjects with PrR (-) tumors enrolled directly into Treatment Period 2.
Groups:
- PrR (+) Subjects: Subjects noted at Screening to have PrR (+) tumors were enrolled into Treatment Period 1 (TP1) receiving Progestin Monotherapy. Subjects noted to have Progressive Disease rolled into Treatment Period 2 (TP2) and received combination therapy of Sodium Cridanimod and Progestin. PrR (+) subjects that had Disease Control or Stable Disease after 24 weeks of Monotherapy treatment were not eligible to participate in TP2 and were discontinued.
- PrR (-) Subjects: Subjects with PrR(-) tumors at screening will be enrolled directly into Treatment Period 2 (TP2) receiving combination therapy of Sodium Cridanimod and Progestin.
Period: Progestin Monotherapy
Arm/Group | PrR (+) Subjects | PrR (-) Subjects
Started | 16 | 0
Completed | 6 | 0
Not Completed | 10 | 0
Not completed — Stable Disease | 8 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Period: Sodium Cridanimod & Progestin Therapy
Arm/Group | PrR (+) Subjects | PrR (-) Subjects
Started | 6 (Subjects with disease progression after progestin monotherapy will roll over into treatment period 2, and receive combination treatment (Sodium Cridanimod and progestin) until documented disease progression.) | 9 (Subjects determined to have PrR negative status from a tumor tissue sample at Screening will enroll directly into Treatment Period 2 and receive combination treatment (Sodium Cridanimod and progestin) until documented disease progression.)
Completed | 0 | 0
Not Completed | 6 | 9
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Disease Progression | 6 | 5
Not completed — Adverse Event | 0 | 2
Period: Safety Follow Up
Arm/Group | PrR (+) Subjects | PrR (-) Subjects
Started | 6 | 9
Completed | 3 | 8
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Transfer of care to hospice | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PrR(-) Subjects: Subjects with PrR(-) tumors at screening will be enrolled directly into Treatment Period 2 (TP2) receiving combination therapy of Sodium Cridanimod and Progestin.
- Total: Total of all reporting groups
Arm/Group | PrR (+) Subjects | PrR(-) Subjects | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 10
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease Control (ODC) as Determined by Radiographic Imaging Measurements
Description: Subjects in the Full Analysis Set (FAS) population will be assessed for ODC. The FAS population includes those subjects all treated in TP2 who either undergo a CT or MRI scan with tumor assessment at 12 weeks (i.e. they have not discontinued treatment prior to 12 weeks) or those who have discontinued TP2 prior to 12 weeks solely due to documented disease progression. Radiographic disease progression and responses will be defined using RECIST 1.1 criteria:
  Control Response(CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions. The appearance of new lesions is also considered progression.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: During TP2 Every 12 weeks, until disease progression up to 24 months
Population: A total of 15 subjects entered Treatment Period 2, which included the 9 subjects who were PrR negative and the 6 subjects who were PrR positive and completed Treatment Period 1, and received treatment with Intramuscular (IM) sodium cridanimod in combination with oral progestin (megestrol acetate). 2 subjects were unevaluable and withdrew prior to meeting criteria for inclusion in FAS population.
Measure: Count of Participants; unit: Participants
Groups:
- Sodium Cridanimod & Progestin Therapy: Sodium Cridanimod and progestin therapy (megestrol acetate) combination
  Sodium Cridanimod: The study will investigate the efficacy of Sodium Cridanimod in conjunction with progestin therapy in a population of subjects with endometrial cancer, who have failed progestin monotherapy or who have been identified as PrR negative.
  progestin therapy: The study will investigate the use of progestin therapy in conjunction with Sodium Cridanimod
Arm/Group | Sodium Cridanimod & Progestin Therapy
Number analyzed (Participants) | 13
Participants
  Progressive Disease | 8
  Stable Disease | 5
  Partial Response | 0
  Control Response | 0

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The best overall response was the best response recorded from the start of Treatment Period 2 until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).To be assigned a status of CR or PR, tumor measurements were confirmed by repeat assessment performed at least four weeks after the criteria for response are first met. Best Overall Response (OR) was determined based on the following combinations of repeat assessments: CR + CR = CR, CR + PR= SD, PD or PR, CR + SD =SD, CR+ PD = SD, CR + NEW= SD, PR + CR= PR, PR + PR= PR, PR+ SD= SD, PR + PD= SD, PR+ NEW = SD.
Time Frame: 24 months
Population: A total of 15 subjects entered Treatment Period 2, which included the 9 subjects who were PrR negative and the 6 subjects who were PrR positive and completed Treatment Period 1, and received treatment with IM sodium cridanimod in combination with oral progestin (megestrol acetate). Four (4) subjects withdrew from the study prior to meeting evaluable criteria for ORR
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Cridanimod & Progestin Therapy
Number analyzed (Participants) | 11
Participants
  Progressive Disease | 8
  Stable Disease | 3
  Control Response | 0
  Partial Response | 0

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progressive Disease was assessed using RECIST Guideline (version 1.1) whereas at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. Progression-free Survival (PFS) was defined as the duration of time from initiation of Treatment Period 2 (Day 0) until disease progression or death from any cause, whichever occurs first. For the purpose of analysis of PFS, subjects with an unknown response were censored.
Time Frame: 24 months
Population: A total of 15 subjects entered Treatment Period 2, which included the 9 subjects who were PrR negative and the 6 subjects who were PrR positive and completed Treatment Period 1, and received treatment with IM sodium cridanimod in combination with oral progestin (megestrol acetate). Four (4) subjects withdrew from the study prior to meeting evaluable criteria for PFS.
Measure: Number; unit: days
Arm/Group | Sodium Cridanimod & Progestin Therapy
Number analyzed (Participants) | 11
days
  001-15-01 | 168
  001-30-01 | 54
  001-39-05 | 85
  001-45-02 | 85
  001-48-01 | 166
  001-01-03 | 31
  001-39-07 | 32
  001-39-08 | 88
  001-43-01 | 60
  001-45-01 | 144
  001-47-03 | 73

4. Secondary Outcome: Duration of Stable Disease
Description: Stable Disease (SD) was assessed using RECIST Guideline (version 1.1) whereas neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Duration of Stable Disease was defined as the duration of time from initiation of Treatment Period 2 (Day 0) until the criteria for disease progression were first met. For the purpose of analysis of Duration of SD, subjects who died before documented progressive disease were censored.
Time Frame: 24 months
Population: A total of 15 subjects entered Treatment Period 2, which included the 9 subjects who were PrR negative and the 6 subjects who were PrR positive and completed Treatment Period 1, and received treatment with IM sodium cridanimod in combination with oral progestin (megestrol acetate). Four (4) subjects withdrew from the study and 8 subjects did not meet the criteria to be evaluable for duration of SD.
Measure: Number; unit: days
Arm/Group | Sodium Cridanimod & Progestin Therapy
Number analyzed (Participants) | 3
days
  001-15-01 | 168
  001-48-01 | 166
  001-45-01 | 144

5. Secondary Outcome: Overall Survival (OS)
Description: Once disease progression was documented in Treatment Period 2, subjects returned for the Safety Follow-up Visit four (4) weeks following the last treatment and continued to be followed for an additional 12-month period for overall survival. Overall Survival (OS) was defined as the duration of time from initiation of Treatment Period 2 (Day 0) until the subject's death from any cause. For the purpose of analysis of OS, if a subject is alive at the date of last contact the subject was censored at that date of contact.
Time Frame: 12 months
Population: Fifteen (15) subjects who participated in Treatment Period 2 were eligible to be followed for OS; however, 4 of these subjects elected to not participate in the Follow-up Period because of withdrawal of consent (3 subjects) or other (1 subject, subject transferred to hospice). For the 11 subjects who participated in the Follow-up Period for OS, the time (in number of days) from the date of discontinuation to the time of death or last contact for survival information ranged from 32 to 457 days.
Measure: Number; unit: days
Arm/Group | Sodium Cridanimod & Progestin Therapy
Number analyzed (Participants) | 11
days
  001-15-01 | 529
  001-30-01 | 411
  001-39-05 | 473
  001-45-02 | 541
  001-48-01 | 490
  001-01-03 | 77
  001-39-07 | 32
  001-39-08 | 394
  001-43-01 | 65
  001-45-01 | 386
  001-47-03 | 438

ADVERSE EVENTS:
Time Frame: The Investigator will assess subjects for Adverse Events (AEs) at each study visit from signing of Informed Consent through the End of Study Visit/Safety Follow-up Visit, an average of 24 months. All AEs observed or reported after the subject has provided informed consent must be recorded in the source data and reported on the eCRF regardless of causal relationship. No AEs will be recorded during the Safety Follow Up Period during which time only Overall Survival Rate is assessed.
Groups:
- Progestin Monotherapy: Treatment Period 1 (Progestin Monotherapy): During Treatment Period 1, all subjects determined to be PrR positive will receive progestin monotherapy, megestrol acetate, for up to 24 weeks. Subjects will have an MRI or CT scan after 12 and 24 weeks of progestin monotherapy, with response to treatment being assessed according to RECIST 1.1 criteria. All subjects that achieve disease control confirmed by tumor assessment after Treatment Period 1, will be ineligible to enter Treatment Period 2. These subjects will be terminated from the trial and treated according to local standards of practice, which may include continued progestin therapy.
- Sodium Cridanimod & Progestin Therapy: Treatment Period 2 (Combination Treatment): All subjects determined to be PrR negative at Screening and those who received at least 4 weeks of progestin monotherapy and who experienced disease progression at the conclusion of Treatment Period 1 will enter Treatment Period 2 of the study. During Treatment Period 2, subjects will receive Sodium Cridanimod in combination with continued progestin treatment, megestrol acetate. Subjects will receive treatment until disease progression as defined according to RECIST 1.1 criteria, with response assessments performed at 12-week intervals.
Arm/Group | Progestin Monotherapy | Sodium Cridanimod & Progestin Therapy
All-Cause Mortality (participants affected / at risk) | 1/16 | 4/15
Serious Adverse Events (participants affected / at risk) | 5/16 | 2/15
Other Adverse Events (participants affected / at risk) | 13/16 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progestin Monotherapy (N=16) | Sodium Cridanimod & Progestin Therapy (N=15)
Thromboembolic event DVT (Vascular disorders) | 1 (1) | 0 (0) — Deep vein thrombosis
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Small intestinal obstruction
bladder infection (Infections and infestations) | 1 (1) | 0 (0) — Cystitis
encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) — Encephalopathy
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hyponatraemia
increase creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) — Renal failure
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary retention
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) — Haematuria
pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) — Pleural effusion
worsening abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) — Abdominal pain
compression atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Atelectasis
difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Dyspnoea
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progestin Monotherapy (N=16) | Sodium Cridanimod & Progestin Therapy (N=15)
dyspnea/dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (2)
fatigue (General disorders) | 5 (5) | 1 (3)
headache (Nervous system disorders) | 2 (2) | 3 (3)
dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
hypertension (Vascular disorders) | 2 (3) | 2 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
dizziness (Nervous system disorders) | 2 (2) | 1 (1)
hot flush (Vascular disorders) | 2 (2) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2)
malignant pleural effusion/pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
peripheral swelling (General disorders) | 1 (1) | 2 (2)
vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
weight increased (Investigations) | 2 (2) | 1 (2)
abdominal pain/abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
asthenia (General disorders) | 2 (2) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 1 (2)
myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was discontinued early due to a change in development strategy and not due safety concern. No safety concerns were noted during the trial. This change in development strategy was the determining factor in the decision to discontinue the study. Because the study was terminated early, the planned analysis was not conducted, as full enrollment was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03077698/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT03077698/SAP_001.pdf
  • Informed Consent Form (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03077698/ICF_002.pdf